CLINICAL TRIAL: NCT06592937
Title: Potentially Modifiable Ventilation Factors Associated With Outcome in Neurocritical Care vs Non-Neurocritical Care Patients - Rational and Protocol for a Patient-Level Analysis of PRoVENT, PRoVENT-iMiC and ENIO (PRIME)
Brief Title: Harmonized and Pooled Database, Named PRIME.
Acronym: PRIME
Status: Completed | Type: Observational
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, Prof. Dr. Marcus J. Schultz, Prof. Dr, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Other Study IDs: PRIME-NEU
Record Dates: First submitted 2024-07-22; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Invasive Ventilation
Keywords: ICU; Invasive ventilation; Respiratory support; Mortality
MeSH Terms: interventions — Noninvasive Ventilation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients receiving invasive ventilation: Patients receiving invasive ventilation, included in PRoVENT, PRoVENT-iMiC, and ENIO
  Interventions: Other: Invasive ventilation

INTERVENTIONS:
Other: Invasive ventilation — Invasive ventilation and respiratory support

SUMMARY:
We merged the dataset of three large observational studies of invasive ventilation in critically ill patients.

DETAILED DESCRIPTION:
PRIME contains the individual patient data of 3 large observational studies of ventilation, 'PRactice of VENTilation in critically ill patients without ARDS' (PRoVENT), 'PRactice of VENTilation in critically ill patients in Middle-income Countries' (PRoVENT-iMiC) and 'Extubation strategies and in neuro-intensive care unit patients and associations with outcomes' (ENIO).

ELIGIBILITY:
All patients in the PRIME database are eligible for participation in the initial analysis presented here. We will exclude patients receiving ventilation fir another reason than acute brain injury.

Ages: 18 Years to 99 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: PROVENT, PROVENT-iMiC and ENIO included various types of patients, receiving ventilation for different reasons. For this first analysis we will select patients receiving invasive ventilation for acute brain injury.
Sampling Method: Non-Probability Sample
Enrollment: 3270 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-07-26 (Actual); Study Completion 2024-07-26 (Actual)

PRIMARY OUTCOMES:
ICU morality | ICU stay, anticipated average 15 days
  any mortality occurred during ICU stay

SECONDARY OUTCOMES:
Mechanical Power | During the first 7 days of invasive ventilation
  All variables or parameters recorded from the ventilator, when the patient is under mechanical ventilation, to calculate the mechanical power (calculated in Joule/minute)

CONTACTS AND LOCATIONS:
Overall Officials: Marcus J Schultz, Prof, Principal Investigator — Amsterdam UMC
Locations (1):
- Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA), Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
Notably, after this initial analysis of PRIME, the database is available for post-hoc analysis.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: After our first pubblication (next six months) and they will remain available for ever
Access Criteria: For this, interested investigators will have to provide a detailed analysis plan, containing a testable hypothesis, clearly described endpoints and an analysis plan. After approval, investigators will be provided with a mock database that will allow them to write an analysis script in R. PROVE network investigators will then run the script on the PRIME database and provide the investigators with the results. Any publication from an additional analysis must follow the rules for publication denoted by the PROVE network
URL: https://www.provenetwork.org/home